CLINICAL TRIAL: NCT06246695
Title: A Study to Evaluate the Effect of Itraconazole and Rifampicin on the Pharmacokinetics of Jaktinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK022
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitor group (Experimental): Jaktinib 100mg, once daily on the 1st and 9th days before meal; Itraconazole 200mg, once daily from the 4th day to the 12th day.
  Interventions: Drug: Jaktinib Hydrochloride Tablets; Drug: Itraconazole capsule
- Inducer group (Experimental): 1. Jaktinib 100mg, once daily on the 1st and 12th days before meal, Rifampicin 600mg, once daily from the 4th day to the 14th day.
  2. Rifampicin 600mg, once daily from the 1th day to the 11th day, Jaktinib 100mg, once daily on the 9st and 25th days before meal.
  Interventions: Drug: Jaktinib Hydrochloride Tablets; Drug: Rifampicin Capsules

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Oral Jaktinib 100 mg for 1 day
  Other Names: Jaktinib
Drug: Itraconazole capsule — Oral Itraconazole 200 mg for 9 day
  Other Names: Itraconazole
  Arms: Inhibitor group
Drug: Rifampicin Capsules — Oral Rifampicin 600 mg for 11 day
  Other Names: Rifampicin
  Arms: Inducer group

SUMMARY:
The primary objective of this study was to assess the effect of rifampicin and itraconazole, on the pharmacokinetics (PK) of Jaktinib in healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers aged between 18 and 45 years old;
* Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 28 (including 19 and 28);
* The participant is in good health and has no history of heart, liver, kidney, digestive tract, nervous system, etc.;

Exclusion Criteria:

* The participant were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 32 Days
  Pharmacokinetics of Jaktinib by assessment of maximum plasma concentration
AUC | Up to 32 Days
  Area under the plasma concentration versus time curve (AUC) of Jaktinib
Adverse Events | Up to 32 Days
  Number of Participants With treatment-related Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No